CLINICAL TRIAL: NCT02780596
Title: Management of Infant Night Wakings in Pediatric Primary Care
Brief Title: Infant Night Wakings in Pediatric Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Sarah Honaker, Assistant Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1506090982; N109471 (Other Grant/Funding Number: Indiana University Health Values Grant)
Record Dates: First submitted 2016-05-16; First posted 2016-05-23 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Insomnia; Night Wakings
Keywords: Infant; Toddler; Primary Care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Items1;3 (Experimental): Caregiver is randomly assigned to receive screening items 1 and 3. Item 1: Does CHILD NAME often wake one or more times during the night? Item 3: Do you think CHILD NAME's sleep is a problem?
  Interventions: Other: Item1; Other: Item3
- Items1;4 (Experimental): Caregiver is randomly assigned to receive screening items 1 and 4. Item 1: Does CHILD NAME often wake one or more times during the night? Item 4: Does you think CHILD NAME has a sleep problem?
  Interventions: Other: Item1; Other: Item4
- Items1;5 (Experimental): Caregiver is randomly assigned to receive screening items 1 and 5. Item 1: Does CHILD NAME often wake one or more times during the night? Item 5: Do you have any concerns about CHILD NAME's sleep?
  Interventions: Other: Item1; Other: Item5
- Items2;3 (Experimental): Caregiver is randomly assigned to receive screening items 2 and 3. Item 2: Does CHILD NAME often wake one or more times per night and does an adult go to him/her? Item 3: Do you think CHILD NAME's sleep is a problem?
  Interventions: Other: Item2; Other: Item3
- Items2;4 (Experimental): Caregiver is randomly assigned to receive screening items 2 and 4. Item 2: Does CHILD NAME often wake one or more times per night and does an adult go to him/her? Item 4: Does you think CHILD NAME has a sleep problem?
  Interventions: Other: Item2; Other: Item4
- Items2;5 (Experimental): Caregiver is randomly assigned to receive screening items 2 and 5. Item 2: Does CHILD NAME often wake one or more times per night and does an adult go to him/her? Item 5: Do you have any concerns about CHILD NAME's sleep?
  Interventions: Other: Item2; Other: Item5
- Items3;5 (Experimental): Caregiver is randomly assigned to receive screening items 3 and 5. Item 3: Do you think CHILD NAME's sleep is a problem? Item 5: Do you have any concerns about CHILD NAME's sleep?
  Interventions: Other: Item3; Other: Item5
- Items4;5 (Experimental): Caregiver is randomly assigned to receive screening items 4 and 5. Item 4: Does you think CHILD NAME has a sleep problem? Item 5: Do you have any concerns about CHILD NAME's sleep?
  Interventions: Other: Item4; Other: Item5

INTERVENTIONS:
Other: Item1 — Does CHILD NAME often wake one or more times during the night?
  Arms: Items1;3; Items1;4; Items1;5
Other: Item2 — Does CHILD NAME often wake one or more times per night, and does and adult go to him/her?
  Arms: Items2;3; Items2;4; Items2;5
Other: Item3 — Do you think CHILD'S SLEEP is a problem?
  Arms: Items1;3; Items2;3; Items3;5
Other: Item4 — Do you think CHILD NAME has a sleep problem?
  Arms: Items1;4; Items2;4; Items4;5
Other: Item5 — Do you have any concerns about CHILD NAME'S sleep?
  Arms: Items1;5; Items2;5; Items3;5; Items4;5

SUMMARY:
This study aims to:

1. identify which single item or combination of two items perform best in identifying problematic infant night wakings and
2. describe current practices by pediatricians in addressing problematic infant night wakings.

Using a novel computer decision support system in several primary care clinics, caregivers accompanying their child to a health visit will be randomly assigned to receive two of five items assessing night wakings and/or sleep problems, followed by a validated questionnaire for infant night wakings. If caregiver responses to the items suggest a possible sleep problem, pediatricians will receive a prompt in the electronic health record identifying a possible infant sleep problem. A sub-sample of caregivers will then be interviewed regarding the content of the visit that day.

DETAILED DESCRIPTION:
Study investigators have developed a novel decision support system for implementing clinical guidelines in pediatric practices. CHICA (Child Health Improvement through Computer Automation) combines three elements:

1. pediatric guidelines encoded in Arden Syntax;
2. a dynamic, scannable paper user interface; and
3. an HL7-compliant interface to existing electronic medical record systems.

The result is a system that both delivers "just-in-time" patient-relevant guidelines to physicians during the clinical encounter and accurately captures structured data from all who interact with it. Preliminary work with CHICA has demonstrated the feasibility of using the system to implement and evaluate clinical guidelines.

Investigators propose to expand CHICA to include surveillance and screening algorithms for problematic infant night wakings. While an eventual aim is to create and test specific management tools for addressing sleep problems, aims of the current study focus on 1) testing items for the identification of sleep disruption, and 2) identifying current management practices in pediatric primary care.

All caregivers of children between the ages of 5 and 20 months presenting to one of five primary care health clinics will be randomly assigned to receive two of five items pertaining to sleep on the prescreening form (PSF) that is currently administered as part of standard clinical care. Parents will have the option to respond "yes" or "no." Regardless of their responses on the pre-screener form, each parent will then receive a form containing ten items from the Infant Sleep Questionnaire (ISQ). Two combinations of items that are similar (Items 1/2 and Items 3/4) will not be presented together, resulting in 8 possible arms or combinations of items.

If a child is identified as possibly having a sleep disturbance (e.g., caregiver answered yes to one or two items), CHICA will prominently display this information on the physician worksheet, viewed during the office visit. The PCP will receive feedback (e.g, "CHILD NAME may have problematic night wakings") via the electronic health record. At this time, providers will not be given additional guidance about how to proceed. At the end of the visit, the provider will be asked to indicate whether or not a sleep problem was confirmed based on their clinical judgment.

A sub-sample of caregivers whose primary care provider (PCP) confirmed a sleep problem will be contacted by phone within two weeks of the clinic visit and asked to complete an exit interview. Caregivers will be asked questions about their child's sleep, the content of the visit with their pediatrician that day (e.g., what the pediatrician recommended), their perceptions of those recommendations, and the outcome of those recommendations if they attempted them. Exit interviews will be conducted on an on-going basis until a sample of 100 has been completed. Up to 600 families may be contacted in order to complete 100 interviews.

Collaborators on this study include the following individuals:

Stephen Downs, MD, Indiana University School of Medicine; Tamara Dugan MS, Indiana University School of Medicine; Amy Schwichtenberg, PhD, Purdue University; and Jodi Mindell, PhD; St. Joseph's University

ELIGIBILITY:
Inclusion Criteria:

* Infant between the ages of 5 and 20 months (at the time of the visit)
* Caregiver responds to questions on the prescreening form in the waiting room
* Infant is a patient at one of five participating primary care health clinics in Indianapolis Indiana.
* For participation in the phone interviews, caregiver speaks English.

Exclusion Criteria:

* None

Ages: 5 Months to 20 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3501 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Problematic infant night wakings (per validated questionnaire) | On the day of each visit to the PCP for the duration of the study (18 months) or until patient no longer meets eligibility (e.g. ages out).
  Identifying the individual item or combination of two items that most strongly predict a positive score on the Infant Sleep Questionnaire

SECONDARY OUTCOMES:
Problematic infant night wakings (per provider clinical judgment) | On the day of each visit to the PCP for the duration of the study (18 months) or until patient no longer meets eligibility (e.g. ages out).
  Identifying the individual item or combination of two items that most strongly predict a provider endorsement of a sleep problem
Night wakings management (per caregiver report) | Within two weeks after the visit to the primary care provider
  Descriptive and qualitative responses from the caregiver phone interview. Variables of interest include 1) caregiver description of provider recommendations to address night wakings; 2) caregiver perception of these recommendations; 3) outcome of the recommended action.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Honaker, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No